CLINICAL TRIAL: NCT00259805
Title: A Pilot Study of the Use of Rituximab in the Treatment of Chronic Focal Encephalitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Kenneth D. Laxer, M.D., Medical Doctor, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPMC-IRB25.102; Genentech CFE-001
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Focal Encephalitis; Rasmussen's Encephalitis
Keywords: encephalitis; epilepsy; Rasmussens; rituximab; autoimmune
MeSH Terms: conditions — Encephalitis; Epilepsy | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV Infusion (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 given as an IV infusion once weekly for four doses

SUMMARY:
The purpose of this study is to assess the safety, tolerability and effectiveness of rituximab in the treatment of chronic focal encephalitis.

DETAILED DESCRIPTION:
Chronic Focal Encephalitis (Rasmussen's Encephalitis) is a condition characterized by a progressive hemiparesis, cognitive decline (including loss of language skills if the language dominant hemisphere is involved) and epileptic seizures that are typically refractory to medical treatment (Rasmussen). Attempts to control the seizures with anticonvulsants are ineffective and the only effective treatment to date is a hemispherectomy (surgical removal of half of the brain). Children with CFE who undergo cortical resections or hemispherectomies demonstrate an inflammatory histopathology consisting of perivascular lymphocytic cuffing, gliosis, neuronal loss, microglial nodules and later laminar necrosis and spongy degeneration

Rituximab is a genetically engineered, chimeric; murine/human monoclonal antibody directed against the CD20 antigen found on the surface of normal and malignant pre-B and mature B cells. It was approved by the FDA in 1997 for the treatment of relapsed or refractory low grade or follicular, CD20+, B-cell non-Hodgkin's lymphoma (NHL). Rituximab binds specifically to the CD20 antigen expressed on the surface of both normal and malignant pre-B and mature B cells. In vitro mechanism of action studies have demonstrated that the Fc portion of Rituximab binds human complement and can lead to cell lysis of the targeted cell through complement-dependent cytotoxicity. Additionally, it has been demonstrated that Rituximab has significant activity in assays of antibody dependent cellular cytotoxicity (Reff et al. 1994). More recently, Rituximab has been shown to induce apoptosis in vitro in DHL-4, a human B cell lymphoma line (Maloney et al. 1997). The relative extent to which these individual mechanisms account for the observed depletion of normal and malignant B cells in vivo is unknown.

While CFE represents only a very small percentage of patients with epilepsy, the devastating progressive nature of the disease with out any adequate treatments, relegates these children to the relentless loss of cognitive and motor skills, and continuing seizures. Recent evidence suggests this condition is immune mediated and includes the development of antibodies directed against various brain components including glutamate receptors (GluR3) (Rogers). Brain samples from patients with CFE have demonstrated immunoreactivity for IgG, C4 C8, and MAC (Andrews and Whitney) and involvement of both B and T-lymphocytes. Evidence supporting a role for clonally expanded B lymphocytes was found by Baranzini . By analyzing the T-cell receptor expression in brain lesions using PCR these investigators also demonstrated the local immune response in CFE included restricted T-cell populations probably expanding from a few precursor T-cells responding to discrete antigenic epitopes (Li). Following demonstration of antibodies directed against brain elements in CFE, a patient was treated with plasma exchange which produced a significant improvement in seizure frequency, cognition and hemiparesis, lending support to the hypothesis that circulating antibodies contribute to the disease pathogenesis. Subsequently attempts to modify this disease by immune modification (plasmaphoresis, steroids, gamma globulin) have demonstrated modest improvements but the improvements have been short-lived and have not affected the natural progression of this disease. This pilot study proposes to directly attack the cells (B-cells) thought to be instrumental in the development of this condition. Should this approach to treating CFE be successful it will have a major impact on these children's lives.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic focal encephalitis
* IgG & IgM levels within normal limits
* Adequate renal function
* Stable anticonvulsant drug regimen

Exclusion Criteria:

* Evidence of significant ongoing medical condition or progressive neurologic condition (other than CFE)
* Previous treatment with rituximab
* History of significant recurrent infections, or ongoing active infection
* Receipt of a live vaccine within 4 weeks prior to treatment
* History of severe allergic reactions to humanized or murine monoclonal antibodies
* History of drug, alcohol or chemical abuse within 6 months
* Concomitant malignancies or previous malignancy
* Use of steroids or immunoglobulins during the 4 weeks prior to treatment
* Hemoglobin <8.5 gm/dL, Platelets < 100,00/mm, AST or ALT >2.5 ULN
* Positive Hepatitis B or C serology
* History of positive HIV

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Rituximab in the treatment of CFE. Adverse and serious adverse events during the study period, reasonably or probably related to Rituximab, will be assessed at each study visit up to 12 months. | 12 months
The natural history of CFE is a progressive deterioration in cortical function; therefore, any evidence of stabilization or improvement in measures of motor function, cognition and/or seizure frequency will be evidence of efficacy and will be assessed at | 12 months

SECONDARY OUTCOMES:
The percentage of patients with a 50% reduction in seizure frequency (responder rate) at 6 months post treatment (as compared to the patient's baseline seizure frequency) will be determined. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Laxer, M.D., Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Baranzini SE, Laxer K, Bollen A, Oksenberg JR. Gene expression analysis reveals altered brain transcription of glutamate receptors and inflammatory genes in a patient with chronic focal (Rasmussen's) encephalitis. J Neuroimmunol. 2002 Jul;128(1-2):9-15. doi: 10.1016/s0165-5728(02)00109-1. PMID 12098505
- [Background] Prayson RA, Frater JL. Rasmussen encephalitis: a clinicopathologic and immunohistochemical study of seven patients. Am J Clin Pathol. 2002 May;117(5):776-82. doi: 10.1309/AD8R-560C-4V11-C5E2. PMID 12090428
- [Background] Baranzini SE, Laxer K, Saketkhoo R, Elkins MK, Parent JM, Mantegazza R, Oksenberg JR. Analysis of antibody gene rearrangement, usage, and specificity in chronic focal encephalitis. Neurology. 2002 Mar 12;58(5):709-16. doi: 10.1212/wnl.58.5.709. PMID 11889232
- [Background] Whitney KD, Andrews PI, McNamara JO. Immunoglobulin G and complement immunoreactivity in the cerebral cortex of patients with Rasmussen's encephalitis. Neurology. 1999 Sep 11;53(4):699-708. doi: 10.1212/wnl.53.4.699. PMID 10489029
- [Background] Prayson RA, Bingaman W, Frater JL, Wyllie E. Histopathologic findings in 37 cases of functional hemispherectomy. Ann Diagn Pathol. 1999 Aug;3(4):205-12. doi: 10.1016/s1092-9134(99)80052-5. PMID 10459046
- [Background] Li Y, Uccelli A, Laxer KD, Jeong MC, Vinters HV, Tourtellotte WW, Hauser SL, Oksenberg JR. Local-clonal expansion of infiltrating T lymphocytes in chronic encephalitis of Rasmussen. J Immunol. 1997 Feb 1;158(3):1428-37. PMID 9013988
- [Background] Hart YM, Cortez M, Andermann F, Hwang P, Fish DR, Dulac O, Silver K, Fejerman N, Cross H, Sherwin A, et al. Medical treatment of Rasmussen's syndrome (chronic encephalitis and epilepsy): effect of high-dose steroids or immunoglobulins in 19 patients. Neurology. 1994 Jun;44(6):1030-6. doi: 10.1212/wnl.44.6.1030. PMID 8208394
- [Background] Rasmussen T. Further observations on the syndrome of chronic encephalitis and epilepsy. Appl Neurophysiol. 1978;41(1-4):1-12. doi: 10.1159/000102395. PMID 103497